CLINICAL TRIAL: NCT05924646
Title: CAlgary SAlt for Postural Orthostatic Tachycardia Syndrome Study
Brief Title: CAlgary SAlt for POTS
Acronym: CASA-POTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB23-0779
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: Sodium; Salt; Treatment
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized cross-over trial with two arms: high salt and normal salt (placebo).
Who Masked: Participant, Investigator
Masking Description: Study participants and investigators will be blinded throughout the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Dietary Salt Plus Additional Salt (Experimental): 6 grams of salt in slow release capsules combined with 6 grams of salt in the diet.
  Interventions: Dietary Supplement: Sodium Chloride Capsules
- Moderate Dietary Salt Alone (Placebo Comparator): 6 grams of microcrystalline cellulose in slow release capsules combined with 6 grams of salt in the diet.
  Interventions: Other: Microcystalline Cellulose Capsules

INTERVENTIONS:
Dietary Supplement: Sodium Chloride Capsules — Table salt in slow release capsules.
  Arms: Moderate Dietary Salt Plus Additional Salt
Other: Microcystalline Cellulose Capsules — Microcrystalline Cellulose Capsules (Placebo)
  Arms: Moderate Dietary Salt Alone

SUMMARY:
Many patients with postural orthostatic tachycardia syndrome (POTS) have decreased plasma volume. Current POTS guidelines recommend ~10 g of salt and 2-3 L of fluid per day. Despite this recommendation, there is no long term data evaluating the use of salt in POTS. This randomized, placebo-controlled cross-over trial will evaluate a high salt diet, compared to a normal salt diet over a period of 3 months. Participants will complete 3 in lab evaluations including autonomic function testing, tilt table testing, blood volume and urine sodium evaluation, plasma catecholamine measurements and and cytokine measurements.

DETAILED DESCRIPTION:
Background and Rationale:

Postural Orthostatic Tachycardia Syndrome (POTS) is a form of autonomic cardiovascular disease, primarily in women, that is often disabling. The investigators and others have found that many patients with postural tachycardia have decreased plasma volume. Current POTS guidelines recommend ~10 g of salt and 2-3 L of fluid per day. In a proof of concept dietary salt study, the investigators recently showed 6 days of a high salt diet (300 mEq/d), compared to a low salt diet, increases plasma volume, reduced standing plasma norepinephrine, and reduced HR. The high salt diet reduced the median orthostatic tachycardia by 14 bpm. Currently there is only evidence showing the benefits of supplemental salt-intake over one week. It is unknown whether the increased blood volume from high dietary salt intake will persist over several weeks, or if an "escape mechanism" will reduce blood volumes back to baseline levels. This longer-term clinical trial of high dietary salt and water will address this "escape mechanism" and ongoing dietary compliance in POTS.

Research Question & Objectives:

Primary Hypothesis: The primary hypothesis is that after 6 weeks of a moderate dietary salt plus additional salt diet, the upright HR will be lower than after 6 weeks on a moderate dietary salt alone diet.

Secondary hypotheses: The secondary hypotheses include:

* Symptoms evaluated using the VOSS symptom score after 6 weeks of a moderate dietary salt plus additional salt diet will be reduced compared to after 6 weeks of a moderate dietary salt alone diet;
* Upright stroke volume after 6 weeks of a moderate dietary salt plus additional salt diet will be increased compared to after 6 weeks of a moderate dietary salt alone diet;
* Blood volume after 6 weeks of a moderate dietary salt plus additional salt diet will be increased compared to after 6 weeks of a moderate dietary salt alone diet;
* Upright plasma catecholamines after 6 weeks of a moderate dietary salt plus additional salt diet will be increased compared to after 6 weeks of a moderate dietary salt alone diet;
* Quality of life after 6 weeks of a moderate dietary salt plus additional salt diet will be increased compared to after 6 weeks of a moderate dietary salt alone diet.

  3. Methods: Interventions: All participants will be instructed to each 5-6 g of salt per day in their diet. In the moderate dietary salt plus additional salt arm, participants will receive blinded capsules that contain 6g of salt per day (12x 500g slow- release capsules). They will take 2g of salt 3 times per day. Participants in the placebo arm will receive blinded capsules that contain 6g of microcrystalline cellulose. Protocol compliance will be assessed with 24h urine sodium.

Randomization: This is a blinded cross-over study. The investigators will randomize patients to start with either salt capsules or placebo. After the 6-week study arm, participants will cross-over to the second study arm.

Study Visit Schedule: The study will consist of three in-house study sessions: a baseline assessment, and an assessment at the end of each study arm: moderate dietary salt plus additional salt and placebo. The baseline visit will serve as a screening visit. Each study session will take place over 1 day in the Autonomic Lab at the University of Calgary. There will also be four 24hr urine sodium collections, and multiple online REDCap surveys.

In-Lab Evaluation: The in-lab evaluation sessions while consist of autonomic function testing including a 10-minute tilt test, blood volume assessment, and supine and standing bloodwork. An IV will be started for the blood work.

Urine Sodium: Participants will complete a 24-hr urine sodium test around the time of each in-lab evaluation, as well as before the 1 week study wash in.

Study Surveys: At each assessment point (baseline and end of each arm), the investigators will send participants a secure REDCap survey link. At the end of the study, participants will also receive a patient experience survey. Participants will receive a total of 4 surveys.

ELIGIBILITY:
Inclusion Criteria:

* Physician Diagnosis of POTS as defined by the CCS Consensus Statement and as follows:
* Sustained, excessive orthostatic tachycardia ≥ 30 bpm within 10 minutes standing.
* Absence of orthostatic hypotension (>20/10 mmHg decrease) within 3 minutes standing.
* Chronic orthostatic symptoms that improve with recumbence.
* Age 18-60 years old.
* Ability to attend the Calgary Autonomic Research Clinic in Calgary.
* Resident of Canada

Exclusion Criteria:

* Overt cause for postural tachycardia (i.e., acute dehydration, thyroid disease)
* Participants with somatization or severe anxiety symptoms will be excluded
* Pregnant (self-reported)
* Underlying causes of tachycardia including acute hypovolemia, endocrinopathy, anemia, anxiety, medication effects, recreational drug effects, and prolonged bedrest.
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies
* Fludrocortisone use (due to effects on renal Na+ handling)
* Patients who have received IV saline in the 2 months preceding the study or who plan to receive it during the course of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Upright Heart Rate | 10 Minutes
  Upright heart rate measured during the tilt table test at the end of the moderate dietary salt plus additional salt arm compared to the tilt table test at the end of the moderate dietary salt alone arm

SECONDARY OUTCOMES:
Vanderbilt Orthostatic Symptom Score (VOSS) | 10 Minutes
  VOSS score measured during the tilt table test at the end of the moderate dietary salt plus additional salt arm compared to the tilt table test at the end of the moderate dietary salt alone arm
Systolic Blood Pressure | 10 Minutes
  Upright systolic blood pressure measured during the tilt table test at the end of the moderate dietary salt plus additional salt arm compared to the tilt table test at the end of the moderate dietary salt alone arm
Diastolic Blood Pressure | 10 minutes
  Upright systolic blood pressure measured during the tilt table test at the end of the moderate dietary salt plus additional salt arm compared to the tilt table test at the end of the moderate dietary salt alone arm
Stroke volume | 10 minutes
  Upright stroke volume measured during the tilt table test at the end of the moderate dietary salt plus additional salt arm compared to the tilt table test at the end of the moderate salt alone arm

OTHER OUTCOMES:
Blood Volume | 1 hour
  Blood volume measured at the end of the moderate dietary salt plus additional salt arm compared to the end of the moderate salt alone arm
Upright Plasma Norepinephrine | 10 minutes
  Upright plasma norepinephrine measured during the tilt table test at the end of the moderate dietary salt plus additional salt arm compared to the tilt table test at the end of the moderate dietary salt arm

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada